CLINICAL TRIAL: NCT07294326
Title: A Prospective, Randomized, Controlled Study Comparing the Efficacy of Intranasal Corticosteroids (INCS) Combined With Intranasal Antihistamines (INAH) and INCS Combined With Oral Antihistamines (OAH) in the Treatment of Moderate to Severe Allergic Rhinitis Symptoms
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China-Japan Union Hospital (Other)
Responsible Party: Principal Investigator, Dongdong Zhu, Department Director, China-Japan Union Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025101109
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Histamine Antagonists; Therapeutics

STUDY DESIGN:
Intervention Model Description: Through prospective exploration of the efficacy of intranasal corticosteroids (INCS) combined with intranasal antihistamines (INAH) and INCS combined with oral antihistamines (OAH) in treating moderate to severe allergic rhinitis symptoms, this study aims to provide evidence-based medical evidence for the standardized treatment of patients with moderate to severe allergic rhinitis accompanied by typical nasal and ocular symptoms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal corticosteroids (INCS) combined with oral antihistamines (OAH) used for treatment (Active Comparator): Intranasal corticosteroids (INCS) combined with oral antihistamines (OAH) used for treatment. Fluticasone propionate nasal spray (Fushuliang) combined with Azlastine hydrochloride tablets (Kedumin), Fluticasone propionate nasal spray (Fushuliang) 1 spray (50 µ g Fluticasone propionate) on each side of the nostril, twice a day, and Azlastine hydrochloride tablets (Kedumin) 2mg once a day, twice a day, once an hour before breakfast, once at night before sleep, for 14 consecutive days.
  Interventions: Drug: Intranasal corticosteroids (INCS) combined with oral antihistamines (OAH) used for treatment
- Intranasal corticosteroids (INCS) combined with nasal antihistamines (INAH) used for treatment (Experimental): Intranasal corticosteroids (INCS) combined with nasal antihistamines (INAH) used for treatment. Azolastine and fluticasone nasal spray (Demins) were selected, and one spray (137 µ g Azolastine Hydrochloride and 50 µ g Fluticasone Propionate) was applied to each nostril twice a day for 14 consecutive days.
  Interventions: Drug: Intranasal corticosteroids (INCS) combined with nasal antihistamines (INAH) used for treatment.

INTERVENTIONS:
Drug: Intranasal corticosteroids (INCS) combined with oral antihistamines (OAH) used for treatment — Intranasal corticosteroids (INCS) combined with oral antihistamines (OAH) used for treatment. Fluticasone propionate nasal spray (Fushuliang) combined with Azlastine hydrochloride tablets (Kedumin), Fluticasone propionate nasal spray (Fushuliang) 1 spray (50 µ g Fluticasone propionate) on each side of the nostril, twice a day, and Azlastine hydrochloride tablets (Kedumin) 2mg once a day, twice a day, once an hour before breakfast, once at night before sleep, for 14 consecutive days.
  Arms: Intranasal corticosteroids (INCS) combined with oral antihistamines (OAH) used for treatment
Drug: Intranasal corticosteroids (INCS) combined with nasal antihistamines (INAH) used for treatment. — Intranasal corticosteroids (INCS) combined with nasal antihistamines (INAH) used for treatment. Azolastine and fluticasone nasal spray (Demins) were selected, and one spray (137 µ g Azolastine Hydrochloride and 50 µ g Fluticasone Propionate) was applied to each nostril twice a day for 14 consecutive days.
  Arms: Intranasal corticosteroids (INCS) combined with nasal antihistamines (INAH) used for treatment

SUMMARY:
Through prospective exploration of the efficacy of intranasal corticosteroids (INCS) combined with intranasal antihistamines (INAH) and INCS combined with oral antihistamines (OAH) in treating moderate to severe allergic rhinitis symptoms, this study aims to provide evidence-based medical evidence for the standardized treatment of patients with moderate to severe allergic rhinitis accompanied by typical nasal and ocular symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 12-75 years old, both male and female are welcome;
2. The diagnostic criteria for moderate to severe allergic rhinitis refer to the "Chinese Guidelines for Diagnosis and Treatment of Allergic Rhinitis (2022, revised edition)", which states: (1) Symptoms: the presence of 2 or more symptoms such as paroxysmal sneezing, watery nasal discharge, nasal itching, and nasal congestion, with symptoms lasting or accumulating for more than 1 hour per day, with symptoms appearing for at least 1 year, a single symptom score (TNSS score standard) of 2 points or more, and a total nasal symptom score (TNSS score standard) of 6 points or more. May be accompanied by eye symptoms, including itching, tearing, redness, and burning sensation. (2) Signs: Pale and edematous nasal mucosa, accompanied by watery nasal secretions (3) Allergen testing: at least one allergen SPT and/or serum specific IgE positive, or nasal provocation test positive. (4) Severe or severe symptoms that have a significant impact on quality of life, including (i) sleep disorders, (ii) disruptions to daily activities, leisure, and/or exercise, (iii) disruptions to learning or work, (iv) anxiety, depression, or restlessness;
3. The enrolled patients reside in Northeast China and meet the follow-up requirements, including Hulunbuir City, Xing'an League, Tongliao City, Chifeng City, and Xilingol League in Heilongjiang Province, Jilin Province, Liaoning Province, and Inner Mongolia Autonomous Region;
4. The subjects voluntarily participated in this study and signed a written informed consent form.

Exclusion Criteria:

1. Patients who are allergic to other excipients such as azelastine hydrochloride, fluticasone propionate, or related drugs;
2. Pregnant women;
3. Patients with arrhythmia, severe organic heart disease, glaucoma, prostate enlargement, active tuberculosis, malignant tumors, systemic immune diseases, or uncontrolled active infections, such as acute upper respiratory tract infections, who cannot be treated with relevant drugs;
4. Other patients who are unwilling to cooperate with treatment or unable to cooperate with follow-up due to serious systemic or mental illnesses;
5. There are certain organic diseases of the nasal cavity, such as benign and malignant tumors of the nasal cavity, chronic sinusitis with nasal polyps, etc;
6. Age<12 years old or>75 years old;
7. Patients who have received allergen specific immunotherapy or biologic therapy within the past 6 months;
8. Those who cannot tolerate serious systemic or local adverse reactions during relevant examinations or specimen collection;
9. Researchers believe that patients who cannot be included in the group.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | Before the start of treatment, on the 3rd, 7th, and 14th day of treatment
  Description: The minimum possible scale value is 0, and the maximum possible scale value is 12. The higher scores mean a worse outcome.
Total Ocular Symptom Score (TOSS) | Before the start of treatment, on the 3rd, 7th, and 14th day of treatment
  The minimum possible scale value is 0, and the maximum possible scale value is 9. The higher scores mean a worse outcome.
Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) | Before the start of treatment, on the 3rd, 7th, and 14th day of treatment
  The minimum possible scale value is 0, and the maximum possible scale value is 168. The higher scores mean a worse outcome.
General Health Status Score (SF36) | Before the start of treatment, on the 3rd, 7th, and 14th day of treatment
  The general health status score of patients is evaluated in nine dimensions: physiological function (PF), physiological function (RP), physical pain (BP), general health status (GH), energy (VT), social function (SF), emotional function (RE), mental health (MH), and health change (HT). Scores for each dimension range from 0 to 100, with higher scores indicating higher quality of life

SECONDARY OUTCOMES:
Endoscopic sinus scoring (Lund-Kennedy) | Before the start of treatment, the 14th day of treatment
blood cell count | Before the start of treatment, the 14th day of treatment
serum IgE level | Before the start of treatment, the 14th day of treatment
nasal secretions IgE level | Before the start of treatment, the 14th day of treatment

IPD SHARING:
Plan to Share IPD: Undecided